CLINICAL TRIAL: NCT01718327
Title: A Phase II Open-label Single Arm Study of Sunitinib in Patients With Advanced Cholangiocarcinoma
Brief Title: A Study of Sunitinib in Patients With Advanced Cholangiocarcinoma
Acronym: SUN-CK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUN-CK D09-2; 2011-000073-30 (EudraCT Number)
Record Dates: First submitted 2012-10-22; First posted 2012-10-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Unresectable and Advanced Cholangiocarcinoma
Keywords: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label, single arm (Experimental): single arm: sunitinib until progresion or unacceptable toxicity
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — sunitinib dose :37.5mg/day
  Other Names: sutent

SUMMARY:
For patients with non-resectable cholangiocarcinoma, gemcitabine with cisplatin is considered as the reference treatment in first line chemotherapy. However, the outcomes of these patients remain limited and therefore more effective drugs are warranted. The context of the disease and current data on sunitinib suggest that sunitinib may have activity in patients with advanced non resectable cholangiocarcinoma.

Thereby, it is proposed to conduct an open label single arm trial aiming evidencing activity of sunitinib in such a patient population.

DETAILED DESCRIPTION:
The primary objective is to evaluate the overall survival of patients with advanced and unresectable cholangiocarcinoma treated continuously by sunitinib as second line at the dose of 37.5 mg per day, after one line of chemotherapy and to determine whether sunitinib deserves further studies in this indication.

The secondary objectives are

* To evaluate the criteria of efficacy
* To evaluate the effects of sunitinib on tumor angiogenesis
* To characterize the safety profile of sunitinib
* To identify markers associated with response to sunitinib

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent given according to ICH/GCP, and local regulation.
2. Histologically or cytologically proven intrahepatic cholangiocarcinoma.
3. Disease that is not amenable to surgery, radiation, or combined modality therapy with curative intent.
4. Gemcitabine with or without platinum pre-treated patients with documented progression
5. Local, locally-advanced or metastatic disease documented as having shown progression on a scan (CT, MRI).
6. Measurable tumor according to RECIST criteria with at least one unidimensionally measurable target lesion
7. No evidence of biliary duct obstruction unless obstruction controlled by local treatment or, in whom the biliary tree can be decompressed by endoscopic or percutaneous stenting with subsequent reduction in bilirubin £ 1.5xULN.
8. Age between 18 and 80 years old
9. Eastern Cooperative Oncology Group (ECOG) Performance Status :0-1
10. Life expectancy ≥ 3 months.
11. Ability to swallow oral compound.
12. No acute toxic effects of previous treatment superior to grade to 1.
13. Laboratory requirements:

    Hematologic: absolute neutrophil count (ANC) 1.5 x 103/mm3, platelets 100 x 103/mm3, hemoglobin 9 g/dl and Hepatic: Bilirubin < 1.5 x upper normal limit (ULN), and alkaline phosphatase (AP) 5xULN. AST and ALT may be 5 x ULN Patients with jaundice Prothrombin time and partial thromboplastin time 1.7 xULN, serum albumin 2.8 g/dl. Renal: Serum creatinine 1.5 xULN , and clearance > 60 ml/min.
14. Normal cardiovascular function
15. Adequate organ function
16. No cardiovascular events during the year prior to study entry
17. Female patients must be surgically sterile or postmenopausal, or must agree to use effective contraception during the period of therapy. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) within 7 days prior to starting study drug. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the investigator or a designated associate
18. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
19. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures
20. Registration in a national health care system (CMU included).

Exclusion Criteria:

1. Hilar cholangiocarcinomas, cholangiocarcinomas located in the gall bladder, hepatic capsule effraction, extrahepatic primary cholangiocarcinoma, carcinoma of the Water ampullum.
2. Prior treatment with other chemotherapy than gemcitabine and/or platinum.
3. Concomitant treatment with any chemotherapy, chemoembolization therapy, immunotherapy, antitumoral hormonotherapy or investigational anticancer agents..
4. Prior treatment with any tyrosine kinase inhibitors or anti-VEGF angiogenic inhibitors.
5. Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri.
6. Treatment with potent CYP3A4 inhibitors and inducers within 7 and 12 days, respectively prior to study drug administration.
7. Pre-existing thyroid abnormality of thyroid function that cannot be maintained in the normal range with medication.
8. Concomitant treatment with therapeutic doses of anticoagulants (low dose warfarin (Coumadin) up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed).
9. Unstable systemic diseases including uncontrolled hypertension (>150/100 mmHg despite optimal medical therapy) or active uncontrolled infections.
10. Drug having proarrhythmic potential (terfenadine, quinidine,procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide and flecainide).
11. Any of the following within the 12 months prior to study drug administration: myocardial infarction, severe/unstable angina, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
12. Abnormal cardiac function with abnormal 12 lead ECG. Ongoing cardiac dysrhythmias of NCI CTC grade2, atrial fibrillation of any grade, or prolongation of the QTc interval to >450 msec for males or >470 msec for females.
13. Symptomatic brain metastases, spinal cord compression, or new evidence of brain or leptomeningeal disease.
14. Current treatment with any other investigational medicinal product.
15. Positive test for human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
16. Pregnancy or breastfeeding.
17. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2016-11-17 (Actual); Study Completion 2016-11-17 (Actual)

PRIMARY OUTCOMES:
Overall survival | time interval from first sunitinib dose to the date of death as a result of any cause assessed up to 3 years
  to evaluate the overall survival of patients with advanced and unresectable cholangiocarcinoma treated continuously by sunitinib as second line at the dose of 37.5 mg per day, after one line of chemotherapy and to determine whether sunitinib deserves further studies in this indication.

SECONDARY OUTCOMES:
To evaluate the criteria of efficacy (PFS, ORR) | time interval from first sunitinib dose to documented disease progression or death due to any cause, assessed up to 3 years after the beginning of the study
  Criteria of efficacy will be determined by:
  * The time to progression under treatment defined as time from first sunitinib dose to documented disease progression or death due to any cause.
  * The objective response rate (ORR) defined as the percentage of all patients who experienced a confirmed complete response (CR) and partial response (PR) based on RECIST criteria. The best overall response, defined as the best response recorded from the start of the treatment until disease progression/recurrence, will be considered.
To evaluate the effects of sunitinib on tumor angiogenesis | Time interval from baseline to the end of treatment, an expected average of 6 months
  The effects of sunitinib on tumor angiogenesis will be determined using the following imaging techniques:
  * Tumor density modification assessed on CT-scan
  * The functional response according to modifications of vascular permeability assessed by either dynamic contrast-enhanced (DCE) magnetic resonance imaging parameters and/or diffusion MRI.
To characterize the safety profile of sunitinib (collection of AEs) | Time interval from study entry to 1 month after last study drug administration, assessed up to 3 years after the beginning of the study, assessed up to 7 months after the beginning of the study
  Safety will be determined in this patient population by the evaluation of adverse events assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events.
  In order to ensure complete safety data collection, all AEs occurring during the study, including any pre- and post-treatment periods required by the protocol must be recorded.
  The period of observation for this study is from signature of informed consent or visit 1 to 1 month after last study drug administration.
  Post-treatment follow up (including assessment/follow-up of adverse events) will be performed every 2 months
To identify markers associated with response to sunitinib | Time interval from baseline to the end of treatment, an expected average of 6 months
  markers

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Faivre, MD/PhD, Principal Investigator — Hôpital Beaujon
Locations (6):
- France (6):
  - Hôpital Beaujon, Clichy
  - Hôpital privé Jean Mermoz, Lyon
  - CHU La Timone, Marseille
  - Hôpital Saint Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Gros L, Bouattour M, Dumont C, Dahan L, Malka D, Tijeras-Raballand A, De Gramont A, Ronot M, Dreyer C, Neuzillet C, Bourget P, Hadengue A, Roldan N, Garcia-Larnicol ML, Chibaudel B, Raymond E, Faivre S. Sunitinib as Second-Line Treatment in Advanced Intrahepatic Cholangiocarcinoma: Results From the SUN-CK GERCOR Phase II Trial. Liver Int. 2025 Aug;45(8):e70196. doi: 10.1111/liv.70196. PMID 40631456
- [Derived] Dreyer C, Sablin MP, Bouattour M, Neuzillet C, Ronot M, Dokmak S, Belghiti J, Guedj N, Paradis V, Raymond E, Faivre S. Disease control with sunitinib in advanced intrahepatic cholangiocarcinoma resistant to gemcitabine-oxaliplatin chemotherapy. World J Hepatol. 2015 Apr 28;7(6):910-5. doi: 10.4254/wjh.v7.i6.910. PMID 25937868